CLINICAL TRIAL: NCT01282528
Title: Ultrasonographic Monitoring of Response to Infliximab in Patients With Rheumatoid Arthritis
Acronym: ULTRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other); First Hospital of China Medical University (Other); Shenzhen People's Hospital (Other); Changhai Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First People's Hospital of Foshan (Other); West China Hospital (Other)
Responsible Party: Yan Zhao, Xiaomei Leng, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMICADEART4011
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Rheumatoid Arthritis; Ultrasonography; Infliximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: infliximab — 3mg/kg, at week 0, 2, 6, 14, 22
  Other Names: Remicade

SUMMARY:
To evaluate the predictive value of clinical, functional (HAQ), laboratory and US variables in relation to disease activity and radiographic outcome in patients with RA who start treatment with Remicade at 24 weeks.

DETAILED DESCRIPTION:
This is an open-lable, single arm study of the ultrasonographic monitoring of response to infliximab in patients with rheumatoid arthritis. Approximately 120 subjects will be enrolled. Subjects will receive infliximab 3mg/kg intravenous infusion at 0, 2, 6 week, and then repeated every 8 weeks until 24 weeks.

The efficacy assessment is observed by ACR response, HAQ, DAS28, sharp scores and US assessment at 0,2，6,14, 22, and 24weeks and ultrosonographic and radiographic assessments are conducted at 0, 6,and 24weeks.

Subjects will be followed for AEs and SAEs up to 8 weeks following the last study treatment administration (see Section 6).

The end of study is defined as the time the last subject completes the 24 weeks visit.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years, male or female and who are capable of providing informed consent, which must be obtained prior to any study-related procedures.
2. Those who have a definitive diagnosis of RA based on the criteria of American College of Rheumatology in 1987 and have moderate to severe disease (DAS28 more than 3.2).
3. Patients using oral corticosteroids, must have been on a stable dose of prednisone 10mg/day or its equivalent for at least 4 weeks prior to screening. If currently not using corticosteroids the patient must have not received corticosteroids for at least 4 weeks prior to screening.
4. Patients using DMARDs, must have been on a stable dose for at least 12 weeks prior to screening. If currently not using DMARDs the patient must have not received DMARDs for at least 12 weeks prior to screening.
5. If using NSAIDs or other analgesics for RA, must be on a stable dose for at least 2 weeks prior to the first administration of study agent.

Exclusion Criteria:

1. Patient who has a known hypersensitivity to human immunoglobulin proteins or other components of infliximab.
2. Patient who suffers from systemic inflammatory disease whose signs and symptoms are expected to affect the evaluation of the study drug.
3. Patient who has a history of receiving infliximab or any other biologics.
4. Patient who has stage IV RA.
5. Patient who has had or is on live viral or bacterial vaccinations within 4 weeks to study entry.
6. Patient who ever suffered from chronic or recurrent infection, including but not limited to: chronic kidney infection, chronic thoracic cavity infection (eg. bronchiectasis), nasosinusitis, recurrent urinary tract infection, open, drain or dermal infected wound.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2010-09

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of treatment with infliximab on synovitis in RA patients using ultrasonography at 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
estimate and visualize the efficacy of treatment with infliximab in RA patients using ultrasonography | 6, 24 weeks
investigate the validity and sensitivity of ultrasonography assessment of joints inflammation in patients with RA compared with sharp scores
3) observe the relationship between ultrasonography assessment and DAS28, ACR20 and sharp scores and other clinical index

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, MD, Principal Investigator — Perking Union Medical College hospital; Xiaomei Leng, MD, Principal Investigator — Perking Union Medical College Hospital
Locations (1):
- Perking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Leng X, Xiao W, Xu Z, Zhu X, Liu Y, Zhao D, Xu H, Chen G, Yu W, Lu J, Wang J, Xia X, Li Y, Zhao Y, Tang H, Shi Y, Bao J, Chen L, Lin L, Zhou L, Zhang H, Zhao Y. Ultrasound7 versus ultrasound12 in monitoring the response to infliximab in patients with rheumatoid arthritis. Clin Rheumatol. 2016 Mar;35(3):587-94. doi: 10.1007/s10067-016-3176-2. Epub 2016 Jan 19. PMID 26781785